CLINICAL TRIAL: NCT01863758
Title: Prospective, Open-label, Multicenter Phase 3b Study to Assess the Safety and Efficacy of Individually Tailored Prophylaxis With Human-cl rhFVIII in Previously Treated Adult Patients With Severe Haemophilia A
Brief Title: Assess the Safety and Efficacy of Individually Tailored Prophylaxis With Human-cl rhFVIII in Patients With Severe Haemophilia A
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Octapharma (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: GENA-21
Record Dates: First submitted 2013-05-23; First posted 2013-05-29 (Estimated); Results first posted 2018-01-30 (Actual); Last update posted 2018-01-30 (Actual); Status verified 2017-07

CONDITIONS: Severe Haemophilia A
MeSH Terms: conditions — Hemophilia A

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Human-cl rhFVIII (Experimental): Up to 60-80 IU/kg of intravenous Human-cl rhFVIII was administered at an individually determined dose and dose interval.
  Interventions: Biological: Human-cl rhFVIII

INTERVENTIONS:
Biological: Human-cl rhFVIII — Human-cl rhFVIII was provided as a freeze-dried concentrate to be reconstituted in water for injection.

SUMMARY:
To compare the number of breakthrough bleeds under tailored prophylaxis with Human cell line recombinant factor FVIII (Human-cl rhFVIII) with the historical bleeding rate from patients who received Human-cl rhFVIII as on demand treatment.

DETAILED DESCRIPTION:
There were 3 phases in this study: (1) An initial pharmacokinetic (PK) assessment in which participants received a single infusion of 60±5 IU/kg of Human-cl rhFVIII; blood samples were collected for 72 hours following the infusion. (2) Prophylactic Treatment-Phase I during which participants received infusions of 30-40 IU/kg of human-cl rhFVIII every other day or 3x/week for 1-3 months. (3) Prophylactic Treatment-Phase II during which the dose and dosing interval were determined individually from data gathered in the initial PK assessment. The maximum dosing interval with a dose of ≤ 60-80 IU/kg that maintains a trough level of ≥ 0.01 IU/mL was determined. Participants were treated for 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Severe haemophilia A (FVIII:C < 1%) according to medical history.
* Male patients ≥ 18 years old.
* Previous treatment with a FVIII concentrate (regular prophylaxis with good compliance or on-demand treatment) for at least 150 exposure days (EDs).
* Good documentation regarding dosing and bleeding frequency in the 6 months preceding study start.
* Immunocompetence (CD4+ count > 200/microliter).
* HIV-negative, if positive, viral load < 200 particles/microliter or < 400,000 copies/mL.
* Freely given written informed consent

Exclusion Criteria:

* Any coagulation disorder other than haemophilia A.
* Present or past FVIII inhibitor activity (> 0.6 Bethesda Unit [BU])
* Severe liver or kidney disease.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2013-08; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (20):
- Medical University Vienna, Vienna, Austria
- Bulgaria (3):
  - University Multiprofile Hospital for Active Treatment, Plovdiv
  - Specialized Hospital for Active Treatment, Sofia
  - Multiprofile Hospital for Active Treatment, Varna
- Germany (2):
  - Vivantes Hospital in Friedrichshain, Berlin
  - SRH Kurpfalzklinik Heidelberg GMBH, Heidelberg
- Hungary (2):
  - Hungarian National Healthcare Center, Budapest
  - University of Debrecen, Medical and Health Science Center, Debrecen
- Poland (4):
  - University Teaching Hospital in Bialystok, Teaching Department of Hematology with a Subdepartment of Vascular Diseases, Bialystok
  - University Clinical Center, Teaching Department of Hematology and Transplantology, Gdansk
  - Nicolaus Copernicus Municipal Specialist Hospital, Department of Hematology, Torun
  - Institute of Hematology and Transfusion Medicine, Depart. of Hemostatic Disorders and Internal Diseases, Warsaw
- Romania (2):
  - Sanador SRL, Bucharest
  - Louis Turcanu Emergency Clinical Children's Hospital, Timișoara
- Slovakia (2):
  - University Hospital Saint Cyril and Metod, Bratislava
  - University Hospital Martin, Department of Hematology and Transfusiology, Martin
- United Kingdom (4):
  - Basingstoke and North Hampshire Hospital, Hemophilia, Hemostasis and Thrombosis Center, Basingstoke
  - Royal London Hospital, Barts and the London Hemophilia Center, London
  - Manchester Royal Infirmary, Department of Clinical Hematology, Manchester
  - Royal Hallamshire Hospital, Sheffield

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Human-cl rhFVIII: Up to 60-80 IU/kg of intravenous human-cl rhFVIII (human cell line recombinant Factor VIII) was administered at an individually determined dose and dose interval.
Period: Pharmacokinetic Assessment
Arm/Group | Human-cl rhFVIII
Started | 66
Completed | 66
Not Completed | 0
Period: Prophylactic Treatment-Phase I
Arm/Group | Human-cl rhFVIII
Started | 66
Completed | 66
Not Completed | 0
Period: Prophylactic Treatment-Phase II
Arm/Group | Human-cl rhFVIII
Started | 66
Completed | 64
Not Completed | 2
Not completed — investigator Error of Early Termination | 1
Not completed — Lost to Follow-up | 1

BASELINE CHARACTERISTICS:
Population: Intent-to-treat/prophylactic/safety population: All participants who received at least 1 dose of Human-cl rhFVIII in Phase II and had any data collected after treatment with Human-cl rhFVIII.
Arm/Group | Human-cl rhFVIII
Number analyzed (Participants) | 66
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 65
  >=65 years | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 66
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 65
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  Austria | 1
  Romania | 9
  Hungary | 4
  Poland | 9
  United Kingdom | 6
  Slovakia | 2
  Bulgaria | 31
  Germany | 4
Age [Mean (Standard Deviation); unit: years] | 33.6 (9.9)
Weight [Mean (Standard Deviation); unit: kg] | 80.5 (19.9)
BMI [Mean (Standard Deviation); unit: kg/m^2] | 25.4 (5.4)
Hemophilia Joint Health Score (HJHS) [Mean (Standard Deviation); unit: Units on a scale] — The HJHS is determined through a physical examination of the 6 joints most affected by hemophilia; the elbows, knees, and ankles. Knees and ankles are assessed on 11 items: Swelling, duration of swelling, muscle atrophy, axial alignment, crepitus on motion, flexion loss, extension loss, instability, joint pain, strength, and gait. Elbows are assessed on 9 of the 11 items (axial alignment and gait are not assessed). Each item is assessed on a scale that ranges from 0-1 to 0-4. The total score can range from 0 to 148, with a higher score indicating a bigger effect of hemophilia.
  Units on a scale | 37.4 (25.3)

OUTCOME MEASURES:

1. Primary Outcome: Annualized Number of Bleeding Episodes (BE) in Phase II
Description: The annualized number of total BEs was calculated for each participant as follows: d*y/t, where y = the number of BEs documented in Phase II, t = the number of treatment periods in days, and d = 365.25, the number of days per year. A bleeding episode (BE) was defined as any BE whether treated or not during Phase II of the study; BEs related to surgery were not included. This study was considered as showing efficacy if the annualized number of BEs was reduced by 50% compared to the number of BEs observed in study GENA-01 where patient where severe Hemophilia A patients were treated on-demand (NCT00989196).
Time Frame: Beginning to the end of Phase II (6 months)
Population: Prophylactic treatment population: All participants who received at least 1 dose of Human-cl rhFVIII in Phase II and had any data collected after treatment with Human-cl rhFVIII.
Measure: Mean (Standard Deviation); unit: Annualized number of bleeding episodes
Arm/Group | Human-cl rhFVIII
Number analyzed (Participants) | 66
Annualized number of bleeding episodes | 3.05 (13.43)
Statistical Analysis 1: Comparison: Human-cl rhFVIII; This study was considered as showing efficacy if the annualized number of bleeding episodes (BE) was reduced by 50% compared to the number of BEs observed in study GENA-01 (NCT00989196); Test type: Superiority or Other; p < 0.05, 2-sided, 1-sample Poisson test; Annualized number of bleeding episodes = 3.13, 95% CI 2-sided [2.56 to 3.80] — The annualized number of bleeding episodes in study GENA-01 was 49.36

2. Secondary Outcome: Annualized Number of Spontaneous Bleeding Episodes (BE) in Phase II
Description: The annualized number of spontaneous BEs was calculated for each participant as follows: d*y/t, where y = the number of spontaneous BEs documented in Phase II, t = the number of treatment periods in days, and d = 365.25, the number of days per year. A spontaneous bleeding episode (BE) was defined as a BE whether treated or not during Phase II of the study. BEs related to surgery and BEs due to trauma or due to other causes were not included.
Time Frame: Beginning to the end of Phase II (6 months)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Annualized number of bleeding episodes
Arm/Group | Human-cl rhFVIII
Number analyzed (Participants) | 66
Annualized number of bleeding episodes | 1.84 (8.81)
Statistical Analysis 1: Comparison: Human-cl rhFVIII; This study was considered as showing efficacy if the annualized number of spontaneous bleeding episodes (BE) was reduced by 50% compared to the number of spontaneous BEs observed in study GENA-01 (NCT00989196); Test type: Superiority or Other; p < 0.05, 2-sided, 1-sample Poisson test; Annualized number of spontaneous BEs = 1.90, 95% CI 2-sided [1.46 to 2.43] — The annualized number of spontaneous bleeding episodes in study GENA-01 was 32.23

3. Secondary Outcome: Annualized Number of Bleeding Episodes (BE) in Phase II in Participants With ≤ 2 Treatments/Week
Description: The annualized number of BEs was calculated for each participant as follows: d*y/t, where y = the number of BEs documented in Phase II, t = the number of treatment periods in days, and d = 365.25, the number of days per year. A bleeding episode (BE) was defined as a BE whether treated or not during Phase II of the study. BEs related to surgery were not included.
Time Frame: Beginning to the end of Phase II (6 months)
Population: Prophylactic treatment population: All participants who received at least 1 dose of Human-cl rhFVIII in Phase II and had any data collected after treatment with Human-cl rhFVIII. Only participants who received ≤ 2 treatments/week were included in the analysis.
Measure: Mean (Standard Deviation); unit: Annualized number of bleeding episodes
Arm/Group | Human-cl rhFVIII
Number analyzed (Participants) | 38
Annualized number of bleeding episodes | 4.1 (17.4)

4. Secondary Outcome: Median Dosing Interval During Individually Tailored Prophylaxis
Description: The median time between 2 prophylactic doses of Human-cl rhFVIII in the prophylactic treatment phase II were determined per patient
Time Frame: Beginning to the end of Phase II (6 months)
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: Hours
Arm/Group | Human-cl rhFVIII
Number analyzed (Participants) | 66
Hours
  Beginning of Phase II | 83.1 [56.2 to 94.4]
  End of Phase II | 83.3 [56.2 to 95.6]

5. Secondary Outcome: Dosage Per Week in Phase II
Description: The mean dosage per week during Phase II of the study are reported.
Time Frame: Beginning to the end of Phase II (6 months)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: IU/kg
Arm/Group | Human-cl rhFVIII
Number analyzed (Participants) | 66
IU/kg | 97.7 (23.1)

ADVERSE EVENTS:
Description: Safety population: All participants who received at least 1 dose of Human-cl rhFVIII.
Groups:
- Human-cl rhFVIII: All subject who received at least one dose of intravenous Human-cl rhFVIII (human cell line recombinant Factor VIII).
Arm/Group | Human-cl rhFVIII
Serious Adverse Events (participants affected / at risk) | 5/66
Other Adverse Events (participants affected / at risk) | 24/66
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Human-cl rhFVIII (N=66)
Haematemesis (Gastrointestinal disorders) | 1 (1)
Fracture of Lower Leg (Injury, poisoning and procedural complications) | 1 (1)
Tenotomy of muculus gastrocnemius medialis (Surgical and medical procedures) | 1 (1)
Appendicitis Acuta (Infections and infestations) | 1 (1)
wound inflammation due to surgery (Infections and infestations) | 1 (1)
Pain of lumbar spine (Musculoskeletal and connective tissue disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Human-cl rhFVIII (N=66)
Nasopharyngitis (Infections and infestations) | 5 (5)
Tonsillitis (Infections and infestations) | 2 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 (4)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2)
Headache (Nervous system disorders) | 5 (5)
Toothache (Gastrointestinal disorders) | 2 (2)
Malaise (General disorders) | 2 (2)
Pyrexia (General disorders) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Octapharma agreements may vary with individual investigators, but will not prohibit any investigator from publishing. Octapharma supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial. Octapharma also reserves the right to review data prior to publishing and provide comments/changes within a certain time period.